CLINICAL TRIAL: NCT06267677
Title: Efficacy of a Specific Complete Formula on Nutritional Status and Coverage of Protein Requirements After Obesity Surgery Compared to the Traditional Progressive Diet: a Prospective Randomized Study
Brief Title: Efficacy of Liquid Versus Powder Protein Supplementation to Optimize Protein Intake After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Violeta Moizé, PhD, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007/3928
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2007-12

CONDITIONS: Body Composition; Obesity; Protein Supplementation; Bariatric Surgery Candidate; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High protein liquid formula (Experimental): Patients allocated in the intervention group (n=15) received 4 high-protein shakes and the corresponding standard vitamin-mineral (VM) supplementation according to our post BS protocol, then progressed towards a diet that combines traditional foods with 2 hLF shakes per day and VM supplementation for 15 days. Over the following 15 days, patients continued to normalize their diet, including a single hLF shake per day and continued with VM supplementation.
  Interventions: Dietary Supplement: High protein liquid formula
- Standard care diet (No Intervention): Patients in the control group (n=35) followed the traditional protocol after bariatric surgery (sCD-group) consisting of a progressive diet with traditional foods, recommendation of 23g/d of protein powder and standard vitamin-mineral supplementation during the first 2 weeks after the surgery. From then on and according to current dietary protocols, the recommendation for protein powder decreases from 23g to 15g up to the end of the study.

INTERVENTIONS:
Dietary Supplement: High protein liquid formula — liquid and high amount of protein
  Arms: High protein liquid formula

SUMMARY:
The goal of this randomized control trial is to compare the effect of a liquid formula rich in nutrients and low in calories (supplement) with the progressive diet with conventional foods that we usually recommend in patients after surgery. The main question it aims to answer is if the addition of a high-protein, volume-controlled nutritional supplement as a fundamental part of the diet during the first two months after surgery will preserve the patient's nutritional status and prevent the appearance of nutritional deficits and associated complications.

Participants will be evaluated at the beginning, at 1 month and at the end of the study (2m) and the following determinations will be made:

* Analytical determination
* Nitrogen balance by determining urea N2 in 24-hour urine
* Anthropometric determinations
* Body composition determined by impedanciometry
* Resting energy expenditure and nutrient oxidation measured by indirect calorimetry.
* Energy, protein and hydration intake.
* Gastrointestinal tolerance through self-registration of symptoms. Researchers will compare the effect of a complete hypocaloric liquid formula group with the usual progressive diet group to see if they achieve the protein intake goal established for patients after obesity surgery, preservation of nutritional status and lean mass during the rapid phase of weight loss and the gastrointestinal tolerance during the first two months after surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients of both sexes between 18 and 65 years of age undergoing bariatric surgery in our center With the ability to understand the objectives and proposals of the study That they agree to participate in the study.

Exclusion Criteria:

Patients who have had perioperative complications and who require an extended hospital stay Patients who after the intervention require some type of artificial nutritional support Patients who have undergone a surgical technique other than BPG.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-01-02 (Actual); Primary Completion 2008-04-18 (Actual); Study Completion 2009-03-06 (Actual)

PRIMARY OUTCOMES:
protein intake | 2 months
  Achieving the protein intake goal established for patients after obesity surgery.
evaluate nutritional deficiencies | 2 months
  Nutritional status and the preservation of lean mass during the rapid phase of weight loss
Tolerance | 2 months
  Gastrointestinal tolerance during the first two months after surgery.

IPD SHARING:
Plan to Share IPD: No